CLINICAL TRIAL: NCT01621828
Title: A Prospective Randomised Controlled Trial of the Impact of Multimedia Information to Reduce Pre-operative Anxiety in Patients Undergoing Major Elective Surgery
Brief Title: Multimedia Information and Pre-operative Anxiety
Acronym: MIPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRO1879
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Anxiety
Keywords: pre-operative anxiety; multimedia information; operating theatre
MeSH Terms: conditions — Anxiety Disorders | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- video (Other): video showing a patient's pathway into the operating room.
  Interventions: Other: video
- leaflet (Other): a written leaflet, about the operating room experience and environment.
  Interventions: Other: leaflet

INTERVENTIONS:
Other: video — a video, showing the patient pathway to and from the Operating Theatre, about the operating room experience and environment.
  Other Names: operating room video
  Arms: video
Other: leaflet — a written leaflet, about the operating room experience and environment.
  Other Names: operating room leaflet
  Arms: leaflet

SUMMARY:
The aim of this study is to investigate a possible reduction in pre-operative anxiety in patients undergoing major elective surgery, by providing multimedia information regarding the patient pathway to and from the Operating Theatre.

DETAILED DESCRIPTION:
To determine whether multimedia information reduces the level of pre-operative anxiety in patients undergoing major elective surgery. To evaluate the efficacy of a video, showing the patient pathway to and from the Operating Theatre, compared with standard information, a written leaflet, about the operating room experience and environment.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing major elective surgery, never previously undergoing surgery as an adult (>18) and admitted to hospital at least one day before the scheduled surgery.

Exclusion Criteria:

* Patients unable to give consent.
* Patients not able to watch the video.
* Patients admitted the same day of the planned surgery.
* Patients not at the first experience of surgery as an adult (>18).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
pre-operative anxiety | two months
  To determine whether multimedia information reduces the level of pre-operative anxiety in patients undergoing major elective surgery. To evaluate the efficacy of a video, showing the patient pathway to and from the Operating Theatre, compared with standard information, a written leaflet, about the operating room experience and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Silvestre, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust Charing Cross Hospital, London, United Kingdom